CLINICAL TRIAL: NCT07101848
Title: A PHASE II, RANDOMIZED TRIAL TO ASSESS MAINTENANCE THERAPY WITH CEMIPLIMAB VERSUS BEST SUPPORTIVE CARE AFTER 1ST LINE PLATINUM-BASED CHEMOTHERAPY IN ADVANCED/RECURRENT VULVAR CANCER
Acronym: BRAVA VULVAR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10021
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Vulvar Cancers
MeSH Terms: conditions — Vulvar Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Cemiplimab maintenance plus best supportive care: cemiplimab 350 mg IV every 3 weeks until week 24, disease progression, unacceptable toxicity or consent withdrawal. Patients who continue to derive clinical benefit on the experimental arm may continue to receive treatment until week 48.
  Interventions: Drug: Cemiplimab
- No intervention (No Intervention): Best supportive care.

INTERVENTIONS:
Drug: Cemiplimab — Cemiplimab maintenance plus best supportive care: cemiplimab 350 mg IV every 3 weeks until week 24, disease progression, unacceptable toxicity or consent withdrawal. Patients who continue to derive clinical benefit on the experimental arm may continue to receive treatment until week 48.
  Arms: Experimental

SUMMARY:
This is a phase II, randomized study that will include 42 participants who have received 4 to 6 cycles of first-line platinum-based chemotherapy for advanced vulvar squamous cell carcinoma (SCC) not amenable to curative surgical treatment (FIGO 2018 stages III-IV - International Federation of Gynecology and Obstetrics) /

recurrent disease, and who have not progressed at the end of these 4 to 6 cycles. Participants eligible for the study will be randomized between 4 and 8 weeks after the last chemotherapy cycle to receive: - Cemiplimab maintenance plus best supportive care: cemiplimab 350 mg IV every 3 weeks until week 24, disease progression, unacceptable toxicity or consent withdrawal. Patients who continue to derive clinical benefit on the experimental arm may continue to receive treatment until week 48. - Best supportive care.

ELIGIBILITY:
Inclusion Criteria:

1) Female participants. 2) At least 18 years old on the day of signing the informed consent. 3) Histologically confirmed diagnosis of vulvar squamous cell carcinoma, clinical stages III-IVA or recurrent disease not amenable to curative-intent therapy, or metastatic disease (stage IVB) - according to FIGO 2018 (International Federation of Gynecology and Obstetrics).4) Measurable disease (as per RECIST v1.1) prior to starting first-line chemotherapy. Lesions located in a previously irradiated area are deemed as measurable if progression has been shown in such lesions. 5) Previous chemotherapy performed in localized disease setting, with curative intent and platinum-based is allowed, provided that the time off this treatment is longer than 6 months. 6) Previous first-line chemotherapy should have been comprised of at least 4 cycles and no more than 6 platinum-based chemotherapy cycles. 7) No evidence of progressive disease after completing first-line chemotherapy (e.g., ongoing complete response (CR), (partial response) PR or stable disease (SD) as per RECIST v1.1 guidelines). 8) An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 or 2.

Exclusion Criteria:

* 1) History of allergy or hypersensitivity to the study drug components. 2) Persisting NCI CTCAE v5.0 Grade > 1 toxicity related to previous therapy; however, Grade ≤ 2 sensory neuropathy and Grade ≤ 2 chronic kidney disease are acceptable. 3) Previous immune therapy with IL-2, IFN-α, or anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-T cytotoxic lymphocyte related to antigen-4 (CTLA-4), or any other antibody or drug specifically targeted to T-cell co-stimulation or immune checkpoint pathways. 4) Untreated or active primary brain tumor, metastases to central nervous system, leptomeningeal disease or spinal cord compression. 5) History of allogenic organ transplant. 6) Ongoing or recent evidence (within 5 years) of significant autoimmune disease requiring treatment with systemic immunosuppressants. 7) History of other primary malignancy within the last 3 years, except locally curable cancers which have been apparently cured, such as skin basal- or squamous-cell cancer, superficial bladder cancer, breast carcinoma in situ or cervical carcinoma in situ. 8) Uncontrolled infection by human immunodeficiency virus, hepatitis B or C infection; or immunodeficiency diagnosis. 9) Have received a live vaccine within 4 weeks of the planned start of the study drug. 10) Have received any previous systemic biological therapy within 5 half-lives of the first study therapy dose.

Exception: participants previously treated with bevacizumab, cetuximab, rituximab or other non-immunomodulating antibodies with half-lives longer than 7 days are allowed after a discussion with the sponsor, if at least 28 days have elapsed since last treatment. 11) Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 42 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From enrollment to 24 weeks
  To assess progression-free survival at week 24 according to the investigator of maintenance cemiplimab after first-line chemotherapy in advanced vulvar squamous cell carcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil